CLINICAL TRIAL: NCT02374918
Title: Bright Light Therapy for Treatment of Sleep Problems Following Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Principal Investigator, William D. Killgore, Principal Investigator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1404301151
Record Dates: First submitted 2014-10-15; First posted 2015-03-02 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Concussion, Mild; Post-Concussion Symptoms; Sleep Problems
Keywords: Mild traumatic brain injury; Concussion; Sleep problems; Brain imaging; fMRI
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- mTBI wavelength-1 bright light (Experimental): 30 minutes daily light exposure for 6 weeks
  Interventions: Device: mTBI wavelength-1 bright light
- mTBI wavelength-2 bright light (Placebo Comparator): 30 minutes daily light exposure for 6 weeks
  Interventions: Device: mTBI wavelength-2 bright light
- HC wavelength-1 bright light (Experimental): 30 minutes of light exposure
  Interventions: Device: HC wavelength-1 bright light
- HC wavelength-2 bright light (Placebo Comparator): 30 minutes of light exposure
  Interventions: Device: HC wavelength-2 bright light

INTERVENTIONS:
Device: mTBI wavelength-1 bright light — 6 weeks of daily light exposure, 30 minutes per morning
  Arms: mTBI wavelength-1 bright light
Device: mTBI wavelength-2 bright light — 6 weeks of daily light exposure, 30 minutes per morning
  Arms: mTBI wavelength-2 bright light
Device: HC wavelength-1 bright light — 30 minutes of light exposure
  Arms: HC wavelength-1 bright light
Device: HC wavelength-2 bright light — 30 minutes of light exposure
  Arms: HC wavelength-2 bright light

SUMMARY:
The purpose of the research study is to understand the effectiveness of a six-week course of light exposure on cognitive functioning, mood, activity, and sleep in people that have suffered a head injury leading to a concussion.

DETAILED DESCRIPTION:
Mild traumatic brain injuries (mTBI) or "concussions" are an increasingly prevalent injury in the investigators society. Patients with post-concussion syndrome have been shown to have deficits on tests of short term memory, divided attention, multi-tasking, information processing speed, and reaction time, as well as alteration in mood and emotional functioning. Many patients have other vague complaints including fatigue, dizziness, irritability, sleep disturbances, and chronic headaches. Furthermore, sleep disruption of one of the most common complaints in patients suffering from traumatic brain injuries, with as many as 40 to 65% of patients with mTBI complaining of insomnia. Sleep problems in these patients are associated with poorer outcome, while resolution of the sleep disturbance is associated with improvement in cognitive functioning.

Despite recent evidence of the correlation between sleep quality and recovery from traumatic brain injury, and the well-established role of sleep in neural plasticity and neurogenesis, there have been virtually no direct studies of the causal effects of sleep on recovery following mTBI. However, it is quite likely that sleep plays a critical role in recovery following brain injury.

A particularly promising non-pharmacologic approach that shows potential in improving/modifying abnormalities of the circadian rhythm and sleep-wake schedule is bright light therapy. For the proposed investigation, the investigators hypothesize that bright light therapy may be helpful in improving the sleep of patients with a recent history of mTBI and may also have other mood elevating effects, both of which should promote positive treatment outcome in these individuals. Bright light therapy may increase the likelihood that they will recover more quickly, benefit more extensively from other forms of therapy, and build emotional and cognitive resilience.

This study will also have a healthy control (HC)/effect localization arm that will assist in identifying and mapping the brain systems before and after light exposure so that researchers may develop further insights into the relationship between concussion, light exposure, sleep, and brain function. This healthy control arm will also provide brain targets for study in the analysis of the Main Study Arm.

ELIGIBILITY:
Inclusion criteria:

* Age range between 18 and 50.
* The primary language of the subjects must be English.
* Subjects have experienced a "concussion" or mTBI within the preceding 18 months, but no sooner that 4 weeks prior to their screening. The occurrence of a concussion or mTBI must be documented by a medical report or other professional witness documentation.
* If documented, Glasgow Coma Scale in the range of 13-15 following the injury.
* Subjects must have complaints of sleep difficulties that emerged or worsened following the most recent head injury.
* At least half of subjects must have evidence of sleep onset insomnia or delayed sleep phase disorder.

Exclusion criteria:

* Any other history of neurological illness, current Diagnostic Statistical Manual (DSM-IV) Axis I disorder, lifetime history of psychotic disorder, or head injury with loss of consciousness > 30 minutes
* Complicating medical conditions that may influence the outcome of neuropsychological assessment or functional imaging (e.g., HIV, brain tumor, etc.)
* Abnormal visual acuity that is not corrected by contact lenses
* Metal within the body, claustrophobia, or other contraindications for neuroimaging
* Less than 9th grade education
* Excess current alcohol use (more than 2 instances of intake of 5+ drinks (men) when or 4+ drinks (women) when drinking in the past two months, and/or on average drinking > 2 drinks per day (men); > 1 drinks per day (women) during the past two months
* History of alcoholism or substance use disorder
* Significant use of illicit drugs
* History of marijuana use within the past 6 weeks and/or use of marijuana before the age of 16.

Subjects who engage in shift-work, night work, or who have substantially desynchronized work-sleep schedules (i.e., sleeping later than 10:00 a.m. more than once a week) will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D Killgore, Ph.D., Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from around the city of Tucson. The first participant was enrolled in December 2014. The Effect Localization Arm completed enrollment in April 2015 and the Treatment Arm completed enrollment in May 2019.
Pre-assignment Details: No pre-assignment criteria were needed after enrollment but before study group assignment for the Effect Localization Arm. For the Treatment Arm, participants went through a screening visit before study group assignment and were excluded based on the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | mTBI Wavelength-1 Bright Light | mTBI Wavelength-2 Bright Light | HC Wavelength-1 Bright Light | HC Wavelength-2 Bright Light
Started | 17 | 18 | 22 | 20
Completed | 14 | 17 | 18 | 18
Not Completed | 3 | 1 | 4 | 2
Not completed — Protocol Violation | 2 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mTBI Wavelength-1 Bright Light | mTBI Wavelength-2 Bright Light | HC Wavelength-1 Bright Light | HC Wavelength-2 Bright Light | Total
Number analyzed (Participants) | 17 | 18 | 18 | 18 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 1 | 2 | 7
  Between 18 and 65 years | 14 | 17 | 17 | 16 | 64
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.53 (8.65) | 26.23 (7.62) | 21.61 (2.86) | 22.28 (4.03) | 23.95 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 9 | 10 | 41
  Male | 5 | 8 | 9 | 8 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 6 | 14
  Not Hispanic or Latino | 15 | 15 | 15 | 12 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 16 | 17 | 15 | 15 | 63
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 18 | 18 | 67
Post-Concussive Symptoms - Rivermead Post-Concussion Symptoms Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Population: The RPCSQ was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  units on a scale
    RPQ3: number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    RPQ3 | 3.3 (3) | 3.5 (2.5) |  |  | 3.4 (2.7)
    RPQ13: number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    RPQ13 | 12.3 (13) | 15.9 (8) |  |  | 14.1 (10.9)
Sleep Quality - PSQI [Mean (Standard Deviation); unit: units on a scale] — Population: The PSQI was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  units on a scale
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 1.44 (0.7) | 1.76 (0.66) |  |  | 1.60 (0.69)
Actigraphy - Sleep Efficiency [Mean (Standard Deviation); unit: Percentage of time asleep] — Population: Actigraphy was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  Percentage of time asleep
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 82.53 (4.83) | 80.98 (4.71) |  |  | 81.73 (4.63)
Actigraphy - Wake After Sleep Onset (WASO) [Mean (Standard Deviation); unit: Minutes] — Population: Actigraphy data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  Minutes
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 11.2 (3.02) | 11.97 (3.23) |  |  | 11.60 (3.06)
RBANS total score (index) [Mean (Standard Deviation); unit: units on a scale] — Population: RBANS data was not collected for the HC wavelength-1 and HC wavelength-2 arms.
  units on a scale
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 88.2 (10) | 96.1 (11.5) |  |  | 92.53 (11.4)
PVT average speed - Run 1 [Mean (Standard Deviation); unit: responses/second] — Population: PVT data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  responses/second
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 3.27 (0.41) | 3.52 (0.35) |  |  | 3.39 (0.39)
PVT average speed - Run 2 [Mean (Standard Deviation); unit: responses/second] — Population: PVT data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  responses/second
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 3.22 (0.51) | 3.45 (0.42) |  |  | 3.33 (0.48)
PVT average speed - Run 3 [Mean (Standard Deviation); unit: responses/second] — Population: PVT data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  responses/second
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 3.17 (0.43) | 3.50 (0.59) |  |  | 3.33 (0.53)
ANAM Code Substitution Learning - thruput score [Mean (Standard Deviation); unit: correct responses/minute] — Population: ANAM data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  correct responses/minute
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 46.78 (14.74) | 55.88 (12.39) |  |  | 51.20 (13.79)
ANAM Procedural Reaction Time - thruput score [Mean (Standard Deviation); unit: correct responses/minute] — Population: ANAM data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  correct responses/minute
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 86.83 (19.55) | 97.06 (19.41) |  |  | 95.26 (17.98)
ANAM Mathematical Processing - thruput score [Mean (Standard Deviation); unit: correct responses/minute] — Population: ANAM data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  correct responses/minute
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 17.89 (8.44) | 21.18 (7.38) |  |  | 19.49 (7.89)
ANAM Matching to Sample - thruput score [Mean (Standard Deviation); unit: correct responses/minute] — Population: ANAM data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  correct responses/minute
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 29.5 (8.05) | 33.29 (11.55) |  |  | 31.34 (9.86)
ANAM Code Substitution delay - thruput score [Mean (Standard Deviation); unit: correct responses/minute] — Population: ANAM data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  correct responses/minute
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 41.06 (13.11) | 52.88 (8.72) |  |  | 46.8 (11.96)
ESS total score [Mean (Standard Deviation); unit: units on a scale] — Population: ESS data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  units on a scale
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 8.72 (3.32) | 8.18 (3.28) |  |  | 8.46 (3.27)
FOSQ Total Score [Mean (Standard Deviation); unit: units on a scale] — Population: FOSQ data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
  units on a scale
    number analyzed (Participants) | 17 | 18 | 0 | 0 | 35
    (all) | 17.10 (2.18) | 15.37 (3.82) |  |  | 14.06 (10.86)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality - Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) subscale measurement that was used is overall sleep quality, which is derived from question 6 on the assessment and uses a Likert scale of 0 to 3. A score of 0 represents "very good" sleep quality (better outcome), while a measurement of 3 represents "very bad" sleep quality (worse outcome).
Time Frame: Post 6-week intervention
Population: The PSQI was not administered to the HC wavelength-2 and HC wavelength-1 arms of this study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 18 | 17
score on a scale | 1.28 (.67) | 1.35 (.7)

2. Primary Outcome: Sleep Quality - Actigraphy Sleep Efficiency
Description: Sleep Efficiency is the overall percentage of time that the participant was scored as sleeping during their night of sleep (range: 0-100%). Higher percentages suggest higher sleep quality and a better outcome.
Time Frame: Post 6-week intervention
Population: Actigraphy data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
Measure: Mean (Standard Deviation); unit: percentage of time asleep
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 18 | 17
percentage of time asleep | 82.57 (4.2) | 83.43 (5.11)

3. Primary Outcome: Sleep Quality - Actigraphy Wake After Sleep Onset
Description: Wake After Sleep Onset (WASO) is how many minutes the participant, during their night of sleep, was determined to be awake after their sleep onset. Sleep onset is defined as a state of at least 2 minutes of uninterrupted sleep. Higher values indicate a worse outcome (range: 1-125 minutes).
Time Frame: Post 6-week intervention
Population: Actigraphy data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 18 | 17
minutes | 11.66 (2.91) | 10.4 (3.32)

4. Primary Outcome: Executive Function Task - Multi-Source Interference Task (MSIT)
Description: Neural activation during functional magnetic resonance imaging (fMRI) measuring executive functioning using the MSIT.
Time Frame: Post 6-week intervention
Population: Data was collected for this measure but was unable to be analyzed due to issues extracting the data from the computer it was stored on. In addition, MSIT data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study 6-weeks after the inital visit.
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Performance on Neuropsychological Assessment - Automated Neuropsychological Assessment Metrics
Description: The Automated Neuropsychological Assessment Metrics (ANAM) is a neuropsychological battery that uses individual tests to measure cognitive efficiency in areas including attention, concentration, reaction time, memory, processing speed, and decision making. Subscale scores are put in terms of a throughput score, which is calculated to be a ratio of correct responses per minute, as a way to measure cognitive efficiency in the participant; as such, the units for the throughput scores would be in terms of correct responses/minute. Higher throughput scores indicate increased levels of cognitive efficiency in the relevant subscale. The throughput score ranges for the ANAM subscales are:
  code substitution learning: 0-147 responses per minute procedural reaction time: 0-151 responses per minute mathematical processing: 0-145 responses per minute matching to sample: 0-97 responses per minute code substitution delayed: 0-155 responses per minute
Time Frame: Post 6-week intervention
Population: ANAM data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
Measure: Mean (Standard Deviation); unit: correct responses/minute
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 18 | 17
correct responses/minute
  ANAM Code substitution learning -thruput score | 51.3 (15.8) | 60.3 (10.8)
  ANAM Procedural Reaction Time - thruput score | 89.8 (19.5) | 101.3 (17.9)
  ANAM Mathematical Processing - thruput score | 18 (8.5) | 22.1 (8.2)
  ANAM Matching to Sample - thruput score | 30.5 (10.1) | 33 (12.2)
  ANAM Code substitution delay-thruput score | 43.3 (14.2) | 56.2 (8.9)

6. Primary Outcome: Performance on Neuropsychological Assessment - Repeatable Battery for the Assessment of Neuropsychological Status
Description: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) uses all of its subscales to calculate the RBANS total score (index). To obtain the RBANS total score (index), the raw scores of the subtests must first be computed into index scores for their relevant subscale (different subtest raw scores feed into specific subscales) using RBANS specific tables that have scaled scores embedded and are normed for the age of the participant. The index scores of each subscale are then summed together to get the Sum of Index Scores, which has a possible range of 200-800. Once the Sum of Index Scores is found, the total score (index) is then found using another RBANS specific table with scaled scores embedded within it. The total score (index) has a possible range of 40-160, with a higher total score (index) is related to a better outcome.
Time Frame: Post 6-week intervention
Population: RBANs data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 18 | 17
units on a scale | 88.5 (10.7) | 97.6 (12.2)

7. Primary Outcome: Performance on Neuropsychological Assessment - Psychomotor Vigilance Task
Description: The Psychomotor Vigilance Task (PVT) is a task that tests alertness by having the participant press a button every time they see a stimulus image appear on a screen. This image is presented at random 2-10 second intervals throughout the entirety of the task. The reaction time (RT) is one of the PVT measurements and is the time, measured in milliseconds, that it takes for the participant to view the stimulus image and then press the button, confirming that they have indeed viewed the stimulus image at that time. The PVT measures speed using the following equation: 1/RT * 1000. The PVT measurement used here is average speed, so all the calculated speeds were then averaged over the entire trial period to obtain the final value for that trial at that time point (post-tx 1,2,3). Since the PVT is a timed measurement of reaction times, lower scores are considered 'better' or indicate an increased level of vigilance.
Time Frame: Post 6-week intervention
Population: PVT data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study 6-weeks after the initial visit.
Measure: Mean (Standard Deviation); unit: responses/minute
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 18 | 17
responses/minute
  PVT average speed - Run 1 - post-tx | 3.3 (0.4) | 3.4 (0.3)
  PVT average speed - Run 2 - post-tx | 3.3 (0.7) | 3.4 (0.4)
  PVT average speed - Run 3 - post-tx | 3.3 (0.6) | 3.4 (0.5)

8. Primary Outcome: Daytime Sleepiness - Epworth Sleepiness Scale
Description: The Epworth Sleepiness Scale (ESS) is an 8-item questionnaire that characterizes the likelihood of the participant 'dozing off' during typical daily activities over their last 2 weeks, and uses a 0-3 point Likert scale, where 0 corresponds to "Would never doze" and 3 corresponds to having a "High chance of dozing" during the activity in question. The ESS score is calculated by adding up all the scores for each question, which means that the ESS score has a range of 0-24, while a higher score indicates that the participant had more issues with daytime sleepiness (worse outcome).
Time Frame: Post 6-week intervention
Population: ESS data was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 18 | 17
units on a scale | 9.33 (3.74) | 6.82 (3.11)

9. Primary Outcome: Daytime Sleepiness - Functional Outcome of Sleep Questionnaire
Description: The Functional Outcome of Sleep Questionnaire (FOSQ) questions 1-26 use a 1-4 (ordinal) likert (1 = "No difficulty" with sleepiness, 4 = "Yes, extreme difficulty" with sleepiness) and the participant also has the option of putting 0 = "I don't do this activity for other reasons".
  FOSQ questions 27-30 use a 1-4 Likert scale where 1 = "Very low" in terms of characterizing the level that sleepiness affects different aspects of their intimate romantic relations, while a 4 = "High" amount of impact on their intimate romantic relations.
  The FOSQ total score measurement is determined by calculating the mean of all 5 subscale scores and then multiplying that value by 5 (range: 0-24). A higher score indicates that the participant had more issues with daytime sleepiness.
Time Frame: Post 6-week intervention
Population: FOSQ was not collected for the HC wavelength-2 and HC wavelength-1 arms of this study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 18 | 17
units on a scale | 16.28 (1.88) | 17.33 (2.39)

10. Primary Outcome: Post-Concussive Symptoms (Rivermead Post-Concussion Symptoms Questionnaire)
Description: The Rivermead Post-Concussion Symptoms Questionnaire (RPCSQ) will be used to assess post-concussive symptoms related to sleep. All questions on the RPCSQ use a 0 to 4 Likert scale concerning the severity of experiencing differing symptoms, where 0 = "not experienced" and 4 = "severe problem". As such, having a higher score is indicative that the participant is having more serious sleep issues related to their head injury. The RPCSQ subscale measurements that were used below are: RPQ3, which is the summed scores from the first 3 questions on the form, with the subscale total ranging from 0-12, and RPQ13, which is the summed scores from questions 4 to 16 on the form, with the subscale total ranging from 0-52. The RPQ3 subscale is associated with earlier symptom clusters of post-concussive symptoms as they relate to sleep disturbances, while the RPQ13 subscale is associated with later symptom clusters of post-concussive symptoms as they relate to sleep disturbances.
Time Frame: Post 6-week intervention
Population: The RPCSQ was not administered to the HC wavelength-2 and HC wavelength-1 arms of this study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Wavelength-2 Bright Light | mTBI Wavelength-1 Bright Light
Number analyzed (Participants) | 18 | 17
score on a scale
  RPQ3 | 3 (2.4) | 2.7 (2.7)
  RPQ13 | 12.8 (11.1) | 11.1 (8.3)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | mTBI Wavelength-1 Bright Light | mTBI Wavelength-2 Bright Light | HC Wavelength-1 Bright Light | HC Wavelength-2 Bright Light
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18 | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT02374918/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT02374918/ICF_001.pdf